CLINICAL TRIAL: NCT04788290
Title: An Observational Study Assessing Effects on Quality of Life, Medication Compliance, Treatment Satisfaction in Patients With Combination Therapy With Raloxifene/Cholecalciferol
Brief Title: An Observational Study Assessing Effects in Patients With Combination Therapy With Raloxifene/Cholecalciferol
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-RAB-OS-01
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Osteoporosis
Keywords: Raloxifene; Cholecalciferol; Osteoporosis; Quality of life
MeSH Terms: conditions — Osteoporosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group(No interventional): Other Name: Observational Rabone D®, Once daily administered per the locally approved product information
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Rabone D®, Once daily administered per the locally approved product information

SUMMARY:
This study examines quality of life and patient satisfaction in postmenopausal women receiving raloxifene to prevent/treat osteoporosis, and vitamin D to reduce risk of fracture using clinical practice data. The purpose of this study is to observe quality of life(QOL), medication compliance and patient satisfaction who got combination therapy with raloxifene/cholecalciferol (raloxifene 60mg + cholecalciferol 800 IU, Rabone D®, Hanmi Pharma, South Korea) for 6 months.

DETAILED DESCRIPTION:
Preventing bone loss is an important concern for women during post-menopausal period. Menopause significantly speeds bone loss and increases the risk for osteoporosis. This study was to investigate the effectiveness on quality of life (QOL), patient satisfaction in postmenopausal women receiving raloxifene/cholecalciferol combination therapy. In addition, we analyzed adverse events to assess the safety profile of this drug.

This study is a multicenter, prospective, non-critical observational study of women receiving raloxifene/cholecalciferol (raloxifene 60mg + cholecalciferol 800 IU, Rabone D®, Hanmi Pharma, South Korea) combination therapy to treat or prevent postmenopausal osteoporosis. Data will be collected from patients receiving routine treatment at about 105 primary, secondary, or tertiary medical institutions in South Korea. Each subject visits the institution according to the protocol that designed the follow-up visits for six months to examine changes in, and factors influencing quality of life (EQ-5D-5L method), patient satisfaction with efficacy and convenience (questionnaire), and safety. This study will approved by the institutions' IRBs and is in compliance with clinical research ethics regulations.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who need to prevent/treat osteoporosis
* Subject who got raloxifene/cholecalciferol combination therapy prescription with confirmation by the investigator's medical decision
* Subjects who can consent voluntarily

Exclusion Criteria:

* Patients for whom use of raloxifene/cholecalciferol combination therapy is prohibited
* Pregnant women, nursing women or child-bearing aged females deemed capable of pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women are at elevated risk of rapid onset osteoporosis, suggesting broad merit in prevention and treatment strategies. This study examines quality of life and patient satisfaction in postmenopausal women receiving raloxifene to prevent/treat osteoporosis, and vitamin D to reduce risk of fracture using clinical practice data.
Sampling Method: Non-Probability Sample
Enrollment: 3907 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
The EuroQol EQ-5D | 6 months
  Change and impact factor of quality of life measured with the EuroQol (EQ-5D)
  EQ-5D-5L is designed to measure health conditions and it consists of 5 questions relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Measuring EQ-5D is performed at each visit.
  The EQ-5D-5L consists of descriptive system with 5 dimensions. Each dimension has 5 levels: No problems(1), Slight problems(2), Moderate problems(3), Severe problems(4), and Extreme problems(5).

SECONDARY OUTCOMES:
Medication compliance (Rate of subjects taking more than 80% of the medication) | 6 months
  This study is to learn more about the relationship between quality of life, patient satisfaction and medication compliance. Measuring medication compliance is performed at each visit. The subjects taking more than 80% are defined as compliance group, and the subjects taking less than 80% are defined as non-compliance group. Medication compliance will be compared between compliance group and non-compliance group.
Treatment satisfaction measured with questionnaire (Patient satisfaction) | 6 months
  This study is to learn more about the relationship between quality of life, patient satisfaction and medication compliance. Measuring patient satisfaction is performed at each visit.
  Treatment satisfaction is measured with 5 satisfaction degrees(Extremely satisfied, Satisfied, Moderate, Dissatisfied, and Extremely dissatisfied).
Evaluation of clinical laboratory changes (BTM(Bone turnover marker) CTX) | 6 months
  The following laboratory test is performed at each visit.
  : CTX (lab unit: e.g. ng/L)
Evaluation of clinical laboratory changes (BTM(Bone turnover marker) NTX) | 6 months
  The following laboratory test is performed at each visit.
  : NTX (lab unit: e.g. nM BCE/mM creatinine)
Evaluation of clinical laboratory changes (BTM(Bone turnover marker) BAP) | 6 months
  The following laboratory test is performed at each visit.
  : BAP (lab unit: e.g. mcg/L)
Evaluation of clinical laboratory changes (BTM(Bone turnover marker) P1NP) | 6 months
  The following laboratory test is performed at each visit.
  : P1NP (lab unit: e.g. μg/L)
Evaluation of clinical laboratory changes (BTM(Bone turnover marker) osteocalcin) | 6 months
  The following laboratory test is performed at each visit.
  : osteocalcin (lab unit: e.g. ng/mL)
Evaluation of clinical laboratory changes (25(OH)D level(25-hydroxyvitamin D level) | 6 months
  The following laboratory test is performed at each visit.
  : 25(OH)D level(25-hydroxyvitamin D level) (lab unit: e.g. ng/mL)
Reason for medication change | 6 months
  Reason for medication(prior-medication to prevent/treat osteoporosis and concomitant medications) change is collected at each visit.
Evaluation of quality of life changes compared with prior medication regimens | 6 months
  This study is to learn more about quality of life changes compared with prior medication regimens. At visit 1, all subjects conduct questionnaire surveys about quality of life. If there are subjects having prior medication regimens for osteoporosis treatment/prevention, these regimens are classified by medication group to compare and evaluate the change in quality of life after taking combination therapy with raloxifene/cholecalciferol. The prior medications are standardized according to ATC(Anatomical Therapeutic Chemical) classification and analyzed based on level 4 and level 5. Change of EQ-5D index according to prior medication regimens is analyzed with average difference of the sum value.
Occurrence and aspect of adverse events(AEs) | 6 months
  After receiving Rabone D®, new adverse events and detailed information are collected at visit 2 and visit 3.

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Jeung KIM, Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No